CLINICAL TRIAL: NCT05482191
Title: Healthy Weight Management Project for Overweight and Obesity Children in Ningbo City
Brief Title: Healthy Weight Management Project for Overweight and Obesity Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NBFH20220667
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Treatment activity on lifestyle interventions will target the dietary and exercise factors of childhood obesity.
  Interventions: Behavioral: Lifestyle intervention
- Usual practice group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — This intervention programme will target the influencing factors of childhood obesity to influence the knowledge, attitude and behaviours of school children. Students in the treatment group will receive the following interventions:
  * Develop and implement school policies related to weight loss
  * Distribute health education materials on diet and exercise to students
  * Carry out student health education courses
  * Diet and exercise instruction by professional nutritionist using internet applet
  * Take part in sports activities that are organized by the sports health teacher during school hours.
  Arms: Treatment group

SUMMARY:
Childhood obesity is a significant public health concern worldwide. In China, childhood obesity has dramatically increased as the economy has grown quickly over the past decades. Nonalcoholic fatty liver disease (NAFLD) is tightly associated with obesity, in China, the prevalence of NAFLD in obesity children is 40.0%，the main interventions for NAFLD are lifestyle interventions. Effective strategies to helping students lose weight and alleviate NAFLD through lifestyle interventions may help promote the physical and mental health of obese students.

This study aimed (1)to assess the effectiveness of the intervention compared with the usual practice in treating childhood overweight and obesity; (2) to determine the sustainability of the treatment in preventing overweight and obesity; (3) to help alleviate or reverse NAFLD in obesity children.

Children with overweight and obesity in six primary schools in Ningbo City, Zhejiang Province will be seleted and randomly divided into two groups: the treatment group and the usual practice group. The participants of the study were students in the third grade of primary school, and the treatment will last for one academic year. This treatment activity on lifestyle interventions will target the dietary and exercise factors of childhood obesity.

ELIGIBILITY:
Inclusion Criteria:

* parents agree and support their children's weight loss, and students and parents have informed consent;
* students in third grade aged 8 and 10 years old;
* students with childhood overweight/obesity defined according to the criteria for Chinese children and adolescents.

Exclusion Criteria:

* medical history of heart disease, hypertension, diabetes, tuberculosis, asthma, hepatitis or nephritis;
* obesity caused by endocrine diseases or side effects of drugs;
* abnormal physical development like dwarfism or gigantism;
* physical deformity such as severe scoliosis, pectus carinatum, limp, obvious O-leg or X-leg;
* inability to participate in school sport activities;
* a loss in weight by vomiting or taking drugs during the past 3 months.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 331 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in body mass index (BMI) | 3 months，9 months , 24 months and 36 months
  * weight and height will be combined to report BMI in kg/m^2
  * caculated by terminal value minus baseline value
change in controlled attenuation parameters (CAP) | 3 months，9 months , 24 months and 36 months
  * CAP will be detected by Fibroscan
  * caculated by terminal value minus baseline value
Change in liver stiffness measurement (LSM) | 3 months，9 months , 24 months and 36 months
  * LSM will be detected by Fibroscan
  * caculated by terminal value minus baseline value

SECONDARY OUTCOMES:
Change in BMI z- score | 3 months，9 months , 24 months and 36 months
  * BMI z- score are measures of relative weight adjusted for child age and sex
  * caculated by terminal value minus baseline value
change in blood glucose | 9 months
  caculated by terminal value minus baseline value
change in blood lipids | 9 months
  * include TC, TG, LDL-C, HDL-C
  * caculated by terminal value minus baseline value
change in fasting insulin | 9 months
  caculated by terminal value minus baseline value
change in body fat percentage | 3 months and 9 months
  caculated by terminal value minus baseline value
change in waist circumference | 3 months，9 months , 24 months and 36 months
  caculated by terminal value minus baseline value
change in weight | 3 months，9 months , 24 months and 36 months
  caculated by terminal value minus baseline value
change in cardiorespiratory endurance test | 3 months，9 months , 24 months and 36 months
  caculated by terminal value minus baseline value
change in ALT(alanine transaminase) | 9 months
  caculated by terminal value minus baseline value

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang PP, Wang YX, Shen FJ, Xing YF, Gu JY, Li XY, Jin H, Jin SF, Xu M, Wang HJ, Wang H, Li L. Lifestyle intervention in children with obesity and nonalcoholic fatty liver disease (NAFLD): study protocol for a randomized controlled trial in Ningbo city (the SCIENT study). Trials. 2024 Mar 20;25(1):196. doi: 10.1186/s13063-024-08046-4. PMID 38504343